CLINICAL TRIAL: NCT03452852
Title: Prospective, Randomized Study of Split Thickness Skin Graft in Wounds on Lower Leg After Compression Therapy With Compression Bandage vs. NPWT
Brief Title: Prospective, RCT of Split Thickness Skin Grafts on Lower Leg After Compression Therapy With Compression Bandage vs. NPWT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Martina Eva Kristiansen, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1603-5
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Skin Cancer
Keywords: Split thickness skin graft; Lower leg; Compression therapy; PICO; Coban 2 lite
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPWT (PICO device) (Other): In this arm, investigators will use the PICO system (Smith and Nephew) for compression therapy after split thickness skin graft of leg ulcers.
  Interventions: Device: PICO
- Compression bandaging (Coban 2 lite) (Other): In this arm, investigators will use the Coban 2 lite compression bandaging for compression therapy after split thickness skin graft of leg ulcers.
  Interventions: Other: Coban 2 lite

INTERVENTIONS:
Device: PICO — NPWT with PICO (Smith and Nephew)
  Arms: NPWT (PICO device)
Other: Coban 2 lite — Compression bandaging with Coban 2 lite
  Arms: Compression bandaging (Coban 2 lite)

SUMMARY:
The single center, prospective, randomized trial includes in total 60 patients. We want to compare two different treatment methods for compression therapy for split thickness skin graft in lower leg. The patients are randomized to compression therapy with NPWT (negative pressure wound therapy) using the device PICO or using the compression bandage with Coban 2 lite.

Primary outcome is complete healing of the skin transplant 30 days postoperatively. Secondary outcomes will be to note frequency of infection, bleeding, loss of transplant etc.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Signed informed consent
* Surgical wound (excision of skin cancer)

Exclusion Criteria:

* Malignant melanoma
* Signs of infection
* Exposed tendon/bone in wound
* Burn/chronic wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Healing of skin graft between the two Methods | 30 days postoperatively
  Numbers of patients with 100 % healing of the split thickness skin graft

SECONDARY OUTCOMES:
Percentage of healing between the two Methods | 30 days postoperatively
  Average healing of the split thickness skin grafts
Evaluation of pain with VAS (Visual analogic scale) | 0, 5-7, 10-14 and 30 days postoperatively
  Pain score as measured by VAS
Level of function | 30 days postoperatively
  Evaluate change in daily function after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Moe Berg, MD, PhD, Principal Investigator — Department of Plastic- and reconstructive surgery, Oslo university hospital - Rikshospitalet, Oslo, Norway
Locations (1):
- Department of Plastic- and Reconstructive Surgery, Oslo university hospital - Rikshospitalet, Oslo, Norway